CLINICAL TRIAL: NCT06857682
Title: Haematological Indices as a Prognostic Predictor Among Patients With Acute on Top of Chronic Liver Cell Failure
Brief Title: Neutrophil to Lymphocyte Ratio and Mean Platelet Volume as a Prognostic Predictor Among Patients With Acute on Top of Chronic Liver Cell Failure
Acronym: ACLF
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa Kamel Khalaf, Dr, Assiut University
Other Study IDs: liver cell failure; Assiut University (Other: Faculty of Medicine)
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute on Top of Chronic Liver Cell Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute on chronic liver failure (ACLF) is a clinical syndrome of sudden hepatic decompensation observed in patients with pre-existing chronic liver disease and associated with one or more extrahepatic organ failures and increased mortality.[1][2][3][4] Regardless of the etiology of chronic liver injury, when a clinician follows the natural history of liver injury, the initial uncomplicated chronic liver disease leads to cirrhosis and, later, the decompensation of liver function with ascites, jaundice, portal hypertension with variceal bleeding, and hepatic encephalopathy. Type-A ACLF is an acute worsening of liver function in a patient with chronic liver disease. Type-B ACLF is when this acute decompensation occurs in patients with cirrhosis, while type-C ACLF is acute worsening of liver function in decompensated cirrhotic.

The etiology of ACLF would be related to a precipitating event in the context of a pre-existing liver condition. Hepatic causes include alcohol-related injury, drug-induced liver injury, viral hepatitis (A, B, C, D, and E), hypoxic injury, or liver surgeries including trans jugular intrahepatic portosystemic shunt (TIPS) placement. Extra-hepatic causes mainly consist of bacterial infections and major surgery. An estimated 40% to 50% of patients are labeled as having an unrecognized precipitating event culminating in ACLF.[5][6][7] The precipitating event has a geographical variation, similar to the etiology of acute liver failure. While acute alcohol injury and bacterial infections are the most common precipitating factor of ACLF in the west; reactivation of chronic hepatitis B, acute hepatitis A, and E infection, along with acute alcohol injury and bacterial infections, are most common in Asia.

* CLF can predict mortality in patient with ACLF and need consideratio for liver transplantation
* Between 24%-40% with cirrhosis develop LCF and admitted into hospital

Grading ACLF helps clinicians assess the prognosis, the usefulness of which has been validated in various studies. ACLF is stratified into 3 grades based on its severity:

Grade-1 ACLF is defined as:

* Single renal failure
* Single liver, coagulation, circulatory, or lung failure that is associated with a serum creatinine level of 1.5 to 1.9 mg/dL and/or hepatic encephalopathy grade 1 or grade 2
* A single brain failure with a serum creatinine level of 1.5 to 1.9 mg/dl Grade-2 ACLF is diagnosed when there are 2 organ failures of any combination. Grade-3 ACLF is diagnosed when there are three or more organ failures of any combination.

The neutrophil-to-lymphocyte ratio (NLR) is an easily accessible biomarker for assessing inflammatory status. It has been shown to be predictive of poor outcome in a variety of diseases, such as cardiovascular disease (8), cancer (9), and postoperative infection (10). In cirrhosis, NLR is a recognized predictor of survival in patients with hepatocarcinoma (11) or hepatitis B virus (HBV) infection, as well as in patients awaiting transplantation (12,13). Moreover, it has been shown that in uncomplicated cirrhosis, higher NLR could predict mortality independently of the model for end-stage liver disease (MELD) and Child-Pugh scores (14).

Aim of the work

* Detecting correlation between lymphocyte/neutrophil ratio and mean platelets volume (MPV)
* Short mortality rate in patients with acute in top of chronic liver cell failure
* Comparison between the predictor different prognostic score and lymphocyte/ neutrophil ratio and mean platelets volume (MPV in patients with acute in top of chronic liver cell failure

DETAILED DESCRIPTION:
Aim of the work

* Detecting correlation between lymphocyte/neutrophil ratio and mean platelets volume (MPV)
* Short mortality rate in patients with acute in top of chronic liver cell failure
* Comparison between the predictor different prognostic score and lymphocyte/ neutrophil ratio and mean platelets volume (MPV in patients with acute in top of chronic liver cell failure

ELIGIBILITY:
Inclusion Criteria:

* Laboratory Confirmation

  * Availability of complete blood count (CBC) with differentials (for NLR calculation: neutrophils/lymphocytes).
  * MPV measured at baseline (preferably before interventions like transfusions or antibiotics).
* Clinical Data Availability

  * Sufficient clinical and biochemical data for prognostic scoring (e.g., MELD, Child-Pugh, CLIF-SOFA).
  * Follow-up data for assessing outcomes (e.g., 30-day mortality, transplant-free survival).
* Age & Consent

  * Adults (typically ≥18 years).
  * Informed consent obtained (if prospective study).

Exclusion Criteria:

* Confounding Hematologic Conditions

  * Active hematologic malignancies (leukemia, lymphoma).
  * Recent blood transfusions (within 48-72 hours, as they may alter NLR/MPV).
  * Known myeloproliferative disorders or bone marrow suppression.
* Recent Infections or Inflammatory Conditions

  * Active non-hepatic infections (e.g., sepsis, pneumonia, HIV) unless ACLF is infection-triggered.
  * Autoimmune diseases (e.g., rheumatoid arthritis, SLE) that may affect NLR.
* Medications Affecting NLR/MPV

  * Recent steroid/immunosuppressant use (modifies WBC counts).
  * Chemotherapy or recent surgery (alters inflammatory markers).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years to 85 years
Study Population: above 18 years below 85 years
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
neutrophil / lymphocyte ratio | 12 Moths from 1/10/2024 - 1/10/2026
  * Detecting correlation between neutrophil / lymphocyte ratio and mean platelets volume (MPV)
  * 30 days and 90 days mortality
  * Liver Transplant free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine - Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
The study is intended to be inside Assiut University and there is no other facility participate into the study

REFERENCES:
- [Result] Patil V, Jain M, Venkataraman J. Paracentesis-induced acute kidney injury in decompensated cirrhosis - prevalence and predictors. Clin Exp Hepatol. 2019 Mar;5(1):55-59. doi: 10.5114/ceh.2019.83157. Epub 2019 Feb 20. PMID 30915407
- [Result] Praktiknjo M, Clees C, Pigliacelli A, Fischer S, Jansen C, Lehmann J, Pohlmann A, Lattanzi B, Krabbe VK, Strassburg CP, Arroyo V, Merli M, Meyer C, Trebicka J. Sarcopenia Is Associated With Development of Acute-on-Chronic Liver Failure in Decompensated Liver Cirrhosis Receiving Transjugular Intrahepatic Portosystemic Shunt. Clin Transl Gastroenterol. 2019 Apr;10(4):e00025. doi: 10.14309/ctg.0000000000000025. PMID 30939488
- [Result] Cai JJ, Wang K, Jiang HQ, Han T. Characteristics, Risk Factors, and Adverse Outcomes of Hyperkalemia in Acute-on-Chronic Liver Failure Patients. Biomed Res Int. 2019 Feb 27;2019:6025726. doi: 10.1155/2019/6025726. eCollection 2019. PMID 30937312